CLINICAL TRIAL: NCT04403737
Title: A Pragmatic Randomized Trial Assessing Efficacy of the Rothman Index
Brief Title: Assessing Efficacy of the Rothman Index
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not started
Sponsor: Yale University (Other)
Collaborators: PeraHealth (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2000027462
Record Dates: First submitted 2020-05-14; First posted 2020-05-27 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Inpatients Who Generate at Least Two Rothman Index Scores

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Usual Care (No Intervention): Patients in the control arm will have a Rothman Index calculated but this will not be visible to providers.
- Intervention (Experimental): Patients in the intervention arm will have a Rothman Index calculated and will be visible to providers. Providers will be given a set of clinician-specific recommended-use protocols that they will be encouraged to follow based on the RI thresholds achieved by patients.
  Interventions: Device: Rothman Index

INTERVENTIONS:
Device: Rothman Index — The Rothman Index score will be calculated and visible to providers. Providers will be encouraged to follow a set of recommended-use protocols in response to different levels of the RI threshold.
  Arms: Intervention

SUMMARY:
This study is designed to assess the efficacy of the Rothman Index in combination with a set of recommended-use protocols to improve rates of mortality and/or rates of discharge to hospice care in hospitalized patients.

DETAILED DESCRIPTION:
The Rothman Index (RI), created by PeraHealth, Inc., is a clinical support system used to recognize the early stages of clinical deterioration. It uses time-updated physiological data (vital signs, lab values, nursing assessments) to calculate a single score that objectively quantifies a patient's condition in real-time. The score is used to detect a patient's declining health and predict risk of decompensation and death. Various risk thresholds exist to describe a patient's status. "Medium" risk is defined by a 30% reduction in a patient's RI score over 24 hours, "high" risk is defined by a 40% drop in the RI score over 12 hours, and "very high" risk" is having a score less than or equal to 20 on the RI. Some institutions have created protocols to be followed by providers when an RI risk threshold is reached (such as triggering rapid response team mobilization), however, there are no standardized protocols shared between hospitals, and none which have been rigorously tested to determine whether they effectively reduce mortality and adverse outcomes.

This is a randomized controlled trial to determine the efficacy of the Rothman Index and an associated set of RI-triggered recommended-use protocol sin improving rates of mortality and/or discharge to hospice care among inpatients of two hospitals within the Yale New Haven Health System. All inpatients admitted to any unit within the study sites who generate at least 2 RI index scores will be automatically enrolled and randomized to either usual care, in which the patient's RI score is calculated but remains unavailable to providers (and available only to the study team), or to the intervention group in which the RI is calculated and visible to providers who will be encouraged to follow recommended protocols appropriate to the RI risk threshold achieved.

The primary outcome is the rates of mortality and/or discharge to hospice care. Secondary outcomes include rates of inpatient mortality, ICU transfer, length of hospital stay, incurred costs, 30 day readmission and mortality rates, and rates of transfer to home.

ELIGIBILITY:
Inclusion Criteria:

* Adults inpatients greater than or equal to 18 years of age
* Admitted to any inpatient unit at two study sites within the Yale New Haven Health System
* Has generated at least 2 Rothman Index scores during the present hospital admission

Exclusion Criteria:

* Prior admission in which patient was randomized
* Patient has opted out of electronic health record consent
* Patient in observation status
* Patient admitted to hospice service

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Mortality and/or discharge to hospice care | Assessed from the date of randomization to the date of the first documented death or discharge to hospice during patient's current hospitalization, up to 365 days
  A composite outcome of mortality and discharge to hospice care as determined by medical record review. Either will be adequate to meet this endpoint.

SECONDARY OUTCOMES:
ICU transfer | Assessed from the date of randomization to the date of first documented ICU transfer during patient's current hospitalization, up to 365 days
  ICU transfer as determined by medical record review.
Length of stay | Assessed as the number of days from the date of randomization to the first documented discharge, up to 365 days
  Patient's length of stay with a start time beginning immediately post-randomization and ending at discharge of the present admission.
Incurred hospital costs | Assessed as costs accrued from the date of randomization to the patient's first documented discharge, up to 365 days
  Hospital costs incurred from post-randomization to discharge, as determined by review of hospital billing records.
Readmission | 30 days post-randomization
  Readmission within 30 days post-randomization as determined by medical record review.
30 day mortality | 30 days post-randomization
  Mortality within 30 days of randomization as determined by medical record review.
Discharge to home | Assessed from the date of randomization to the date of the first document discharge to home, up to 365 days
  As determined by medical record review

CONTACTS AND LOCATIONS:
Overall Officials: Francis P Wilson, MD MSCE, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Greenwich Hospital, Greenwich, Connecticut
  - Lawrence + Memorial Hospital, New London, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data underlying results for publication will be made available upon publication of results.
Supporting Information: Study Protocol, SAP
Time Frame: After publication of results; indefinitely.